CLINICAL TRIAL: NCT06112197
Title: Study of Visceral Fat in Type 2diabetic Patients and Its Relation to Microvascular Complications
Brief Title: Study of Visceral Fat in type2diabetic Patients and Its Relation to Microvascular Complications
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Soliman, Ass.lecturer of internal medicine, Sohag University
Other Study IDs: Soh-Med-23-10-13MD
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Visceral Fat; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study the correlation between METS IR and visceral fat in type 2 diabetes and its relation to microvascular complication

DETAILED DESCRIPTION:
The Metabolic Score for Insulin Resistance (METS-IR) is a metabolic index developed with the aim to quantify peripheral insulin sensitivity in humans; it was first described under the name METS-IR by Bello-Chavolla et al in 2018. It was developed by the Metabolic Research Disease Unit at the Institute National de Ciencias Médicas Salvador Zubirán and validated against the euglycemic hyperinsulinemic clamp and the frequently-sampled intravenous glucose tolerance test in Mexican population.It is a non-insulin-based alternative to insulin-based methods to quantify peripheral insulin sensitivity and an alternative to the Homeostatic Model Assessment (HOMA-IR) and the quantitative insulin sensitivity check index (QUICKI).

Very limited research correlate between visceral obesity and microvascular complications in type 2 diabetic patients and how can the metabolic score for insulin resistance predict visceral obesity and microvascular complications in type2 diabetic patients. In this study the investigators will search for these correlations.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years Both male and female subjects Subjects capable of giving consent and voluntarily willing to participate in the study

Exclusion Criteria:

* Chronic kidney disease patients Any nondiabetic nephropathy patients Patients affected by hypertension Patients affected by ocular disorders Neuropathies of other etiologies like chronic liver disease patients, alcoholics, or drug addicts Critically ill patients of type 2 diabetes mellitus Patients who have not given consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of T2DM, either newly diagnosed or previously diagnosed and on treatment with antidiabetic oral hypoglycemic agents or insulin and attending diabetes OPD or admitted to the Medicine Department, were taken as cases. Age- and gender-matched nondiabetic people admitted to the Medicine Department were taken as control subjects. Both these groups will be interviewed, examined, investigated, and included in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-05 (Estimated); Primary Completion 2025-01-05 (Estimated); Study Completion 2025-06-05 (Estimated)

PRIMARY OUTCOMES:
correlation between METS IR and visceral fat in type 2 diabetes | one year
  Study the cor relation between METS IR and visceral fat in type 2 diabetes and its relation to microvascular complication

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud soliman, Study Director — Sohag University
Locations (1):
- Mahmoud Soliman, Sohag, Egypt